CLINICAL TRIAL: NCT04314466
Title: The Effects of Early-life Environmental and Behavioral Factors on Child Growth and Development
Acronym: SSBC
Status: Completed | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Sijia Gu, Principal Investigator, Shanghai Jiao Tong University School of Medicine
Other Study IDs: SCMCIRB-2012033
Record Dates: First submitted 2020-03-11; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Child Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — child： 20ml cord blood and a piece of placenta mother： 15ml venous blood father： 15ml venous blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Shanghai Sleep Birth Cohort Study (SSBC) is a prospective observational study investigating the sleep condition of women in their third trimester and children from the age of 42 days to 6 years. Both subjective and objective tools were used to assess different sleep characteristics, including sleep duration, sleep rhythm and sleep quality. From August 2012 to June 2013, total 277 pregnant women from the eastern division of Renji Hospital in Pudong New Area, Shanghai were included in the study. Demographic information, physical examination, developmental and psychiatric assessment, diet and physical activity, as well as biological samples were collected for further analysis. Main findings of the current study showed the effect of sleep disturbances during the third trimester on emotional regulation and the influence of different sleep characteristics on children's social-emotional development

ELIGIBILITY:
Inclusion Criteria:

* Long-term resident in Shanghai, and no relocation plan for 2 years
* Ultrasonography indicated singleton pregnancy at 34-36 weeks
* Willingness to participate in the study and engage in the follow-up at the specified time
* Neonates were included if they were partus maturus

Exclusion Criteria:

* Preterm labor symptoms during pregnancy
* Gestational hypertension or gestational diabetes mellitus
* Heart, liver, and kidney disease
* Apgar score was 7 or below at 1 minute or 5 minutes with history of asphyxia at birth

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The prospective cohort study was conducted in the eastern division of the Renji Hospital and Shanghai Children's Medical Center in Pudong New Area, Shanghai, which aimed to explore how the perinatal and early life environmental and behavioral factors affect early child growth and development in a longitudinal and prospective mother-child cohort.
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2012-05-20 (Actual); Primary Completion 2013-09-12 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Maternal sleep measured by Pittsburgh Sleep Quality Index(PSQI) | changes from baseline,3 month, 6month, 9month, 12month, 18month, 24 month,36month,48month follow-up
  The PSQI total score represents the sum of component scores for subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medicine, and daytime dysfunction. A PSQI score >5 defined poor sleep quality. Higher scores implied lower sleep quality or more severe sleep disturbance.
Maternal sleep measured by Actiwatch | baseline
  Sleep assessment was a major part of the study. A 7-day assessment of mothers' sleep quality was conducted during the third trimester by using Actiwatch (Respironics, Inc.1001, Actiwatch 2) and sleep diary. Actiwatch is a sleep assessment system based on monitoring individual activity whose evaluation point is based on the sleep diary.
Children sleep measured by Actiwatch | changes from 3 month, 6month, 9month, 12month, 18month, 24 month,36month,48month,72month follow-up
  Sleep assessment was a major part of the study. A 7-day assessment of mothers' sleep quality was conducted during the third trimester by using Actiwatch (Respironics, Inc.1001, Actiwatch 2) and sleep diary. Actiwatch is a sleep assessment system based on monitoring individual activity whose evaluation point is based on the sleep diary.
Children sleep measured by Brief Infant Sleep Questionnaire(BISQ) | changes from birth, 42days,3 month, 6month, 9month, 12month, 18month, 24 month,36month follow-up
  Infant sleep problems reported by the mother and according to Brief Infant Sleep Questionnaire (BISQ). It is not a scale. The variables of the questionnaire included 1) nocturnal sleep duration (between the hours of 7 pm and 7 am); 2) daytime sleep duration (between the hours of 7 am and 7 pm); 3) number of night wakenings; 4) duration of wakefulness during the night hours (10 pm to 6 am); 5) nocturnal sleep-onset time (the time when the child falls asleep for the night); 6) settling time (latency to falling asleep for the night); 7) method of falling asleep; 8) location of sleep; 9) preferred body position; 10) age of child; 11) gender of child; 12) birth order; and 13) role of the responder who completed the BISQ. If the child woke up more than 3 times per night, spent more than 1 hour in wakefulness during the night, or spent less than 9 hours in sleep (day and night), then they were considered as poor sleepers.
Children sleep measured by Children's Sleep Habits Questionnaire (CHSQ) | changes from 48month, 72month follow-up
  Children's Sleep Habits Questionnaire (CHSQ) Sleep onset and wake up time in the past weekdays and weekends were collected from a parent reported Children Sleep Habits Questionnaire23 and sleep duration in weekdays and weekends was calculated separately. Daily average sleep duration was calculated using the formula: ([weekday sleep duration×5] + [weekend sleep duration×2])/7.
Children weight | changes from birth,42days,3 month, 6month, 9month, 12month, 18month, 24 month,36month,48month,72month follow-up
  Child weight were obtained at each visit. Weight was measured using calibrated scales (birth to 24 months, Seca 335, Hamburg, Germany) and electronic personal scale (3-4 years, Seca 877, Hamburg, Germany).
Children length/height | changes from birth,42days,3 month, 6month, 9month, 12month, 18month, 24 month,36month,48month,72month follow-up
  Child length/height were obtained at each visit.Recumbent length (birth to 24 months) was measured from the top of the head to the soles of feet using the same calibrated scale as weight. Standing height (2-4 years) was measured using a stadiometer (Seca 206, Hamburg, Germany) from the top of children's head to his or her heels.
Social-emotion | changes from 36month,48month,72month follow-up
  The Strengths and Difficulties Questionnaire (SDQ) we use in this survey is a short screening questionnaire covering the current difficulties in social psychology (i.e. emotional symptoms, conduct problems, hyperactivity-inattention, peer problems), and personal strengths (i.e. prosocial behavior). High SDQ score is associated with an increase in psychiatric risk, on the opposite, prosocial behavior score is positive with prosocial behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai children's medicial center affiliated shanghai jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China